CLINICAL TRIAL: NCT07008846
Title: Efficacy of Tofacitinib, Methotrexate Combination Therapy Versus Upadacitinib, Methotrexate Combination Therapy in Moderate to Severe Rheumatoid Arthritis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Md Anisul Islam, Director, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 5454
Record Dates: First submitted 2025-05-11; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Moderate to Severe Rheumatoid Arthritis
MeSH Terms: interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Efficacy of upadacitinib, methotrexate combination therapy versus tofacitinib, methotrexate combinat (Experimental)
  Interventions: Drug: To see the efficacy of Upadacitinib, Methotrexate versus Tofacitinib, Methotrexate in moderate to severe Rheumatoid arthritis

INTERVENTIONS:
Drug: To see the efficacy of Upadacitinib, Methotrexate versus Tofacitinib, Methotrexate in moderate to severe Rheumatoid arthritis — This intervention is open label. Both patient and investigator will know about the intervention. Participants are allocated according to block randomization. Total two groups with each contain 48 patients. One group will be given Tofacitinib, Methotrexate and another group will be given Upadacitinib, Methotrexate

SUMMARY:
The aim of this study is to assess the efficacy of upadacitinib, methotrexate combination therapy in comparison to tofacitinib, methotrexate combination therapy in moderate to severe RA patients. This study will guide us to treat RA patients with inadequate response to methotrexate more effectively

ELIGIBILITY:
Inclusion Criteria:

- 1.Patients of both gender (age ≥18 years). 2.Patients fulfill the ACR/EULAR 2010 classification criteria for rheumatoid arthritis.

3.Patients with DAS-28 CRP >3.2 despite optimum dose and duration of methotrexate (20-25 mg/week for minimum one month).

Exclusion Criteria:

* 1.Recent or concurrent infection

  2.Active or latent tuberculosis

  3. Hemoglobin (Hb) < 8 g/dl 4. White blood cell count < 4000/ micro L, Neutrophil count < 1000/ micro L, Platelet count < 100000/mm3 5. Live vaccines (rota virus, varicella, yellow fever) within 3 months prior to the first dose 6. Child-Pugh Class -C 7. Pregnant or planned for pregnancy and breastfeeding females of child-bearing potential 8. Evidence or history of malignancy, with the exception of adequately treated or excised non-metastatic basal or squamous cell cancer of the skin or cervical carcinoma in situ 9. New York Heart Association Class III and IV congestive heart failure 10. Previous history of thromboembolism, deep venous thrombosis, stroke, IHD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
DAS28-CRP | Outcome 1:"Disease Activity Score 28 CRP (DAS28-CRP) at week 4" Outcome 2:"Disease Activity Score 28 CRP (DAS28-CRP) at week 12" Outcome 3:"Disease Activity Score 28 CRP (DAS28-CRP) at week 24"
  Number of Participants with Low disease activity or Remission as Assessed by DAS28-CRP, Change from Baseline in Pain Scores on the Visual Analog Scale at 24Weeks).

CONTACTS AND LOCATIONS:
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Shahbag, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided